CLINICAL TRIAL: NCT02076971
Title: A Multicenter Prospective Observational Study to Evaluate Cytomegalovirus (CMV)-Specific Response Measured by QuantiFeron® and Overall Immunologic Response Measured by ImmuKnow® in Lung Transplant Patients With CMV-positive Serology (R+) Prior to Transplant and Its Involvement in the Development of CMV Infection
Brief Title: Cytomegalovirus-Specific Response Measured by QuantiFeron® and Overall Immunologic Response Measured by ImmuKnow® in Lung Transplant Patients CMV-positive
Acronym: REIVI
Status: Completed | Type: Observational
Sponsor: Fundacio Catalana de Pneumologia (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Principal Investigator, Victor Monforte, Hospital Vall d'Hebron, Fundacio Catalana de Pneumologia
Other Study IDs: FUN-CMV-2013-01
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Cytomegalovirus Infections
Keywords: Lung transplant; Quantiferon; Immuknow
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the sensitivity and specificity of QuantiFeron® and ImmuKnow® in combination for early detection of patients who will develop CMV infection in lung transplant patients with CMV-positive serology (R+) prior to transplant.

DETAILED DESCRIPTION:
The secondary objectives of the study are:

* To evaluate Cytomegalovirus (CMV)-specific immune response measured by QuantiFeron®.
* To evaluate overall immune response measured by ImmuKnow®.
* To study the course of QuantiFeron® and ImmuKnow®over the follow-up period.
* To correlate levels of ImmuKnow® and QuantiFeron®.
* To evaluate the relationship between levels and doses of immunosuppressants and their relationship to degree of overall immunosuppression (ImmuKnow®).
* To evaluate the relationship between infections, immunological complications and degree of overall immunosuppression (ImmuKnow®).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Men or women who have received a lung transplant.
* CMV-seropositive patients (R+).
* Patients who have been informed of the study procedures and have signed the informed consent form.
* Over 3 months posttransplant.

Exclusion Criteria:

* Patients who are not expected to be able to be followed during the first 12 months posttransplant.
* Patient participation in another clinical trial or study will not be a criterion for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CMV-positive (R+) lung transplant patients
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quantification of interferon-γ produced by specific CD8+ (cluster of differentiation 8) T cells after ex-vivo stimulation with various CMV epitopes using the commercial assay QuantiFeron®- CMV | up to 12 months from transplant
  Quantiferon® is assessed multiple times and it will be considered positive when first positive test is assessed.
Measurement of overall immune response by determination of the activity of CD4+ (cluster of differentiation 4) T cells | up to 12 months from transplant
  InmunKnow® is assessed multiple times and it will be considered positive when first positive test is assessed.
Quantification of CMV viral replication in blood measured by PCR (polymerase chain reaction) | up to 12 months from transplant
  PCR is assessed multiple times and it will be considered positive when first positive test is assessed.

SECONDARY OUTCOMES:
Measurement of immunosuppressive drugs: Blood levels of calcineurin inhibitors (tacrolimus or cyclosporine). Mycophenolate (or equivalent) dose and corticosteroid doses. | up to 12 months from transplant
Complete blood count (WBC count) and routine biochemistry | up to 12 months from transplant
Determination of glomerular filtration rate | up to 12 months from transplant
Course of graft function by measuring GFR (glomerular filtration rate) | up to 12 months from transplant
Complications since last visit: Infections, rejection episodes, chronic graft dysfunction, other complications | up to 12 months from transplant
CMV prophylaxis, drug and dosage. Serious Adverse events related or no related to the drug | up to 12 months from transplant
Follow-up loss/death (if it occurs) | up to 12 months from transplant

CONTACTS AND LOCATIONS:
Overall Officials: Victor Monforte, MD, Study Chair — Hospital Vall d'Hebron; Piedad Ussetti, MD, Study Chair — Hospital Puerta de Hierro; Susana Gómez, MD, Study Chair — Hospital Vall d'Hebron Laboratory; Victor Monforte, MD, Principal Investigator — Hospital Vall d'Hebrón; Piedad Ussetti, MD, Principal Investigator — Hospital Puerta Hierro; Francisco Santos, MD, Principal Investigator — Hospital Reina Sofía; José Cifrián, MD, Principal Investigator — Hospital Marqués de Valdecilla; José M Borro, MD, Principal Investigator — Hospital Universitario A Coruña; Virginia Pérez, MD, Principal Investigator — Hospital 12 de Octubre; Amparo Solé, MD, Principal Investigator — Hospital Universitario La Fe
Locations (7):
- Spain (7):
  - Hospital Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario y Politécnico la Fe, Valencia, Valencia
  - Hospital Vall d'Hebrón, Barcelona